CLINICAL TRIAL: NCT06100367
Title: 11C-Metomidate PET/CT for Endocrine Hypertension and Characterisation of Adrenal Tumours
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Collaborators: National University Health System, Singapore (Other); Clinical Imaging Research Centre (Unknown); Singapore General Hospital (Other); Tan Tock Seng Hospital (Other); Khoo Teck Puat Hospital (Other); Ng Teng Fong General Hospital (Other); Sengkang General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA_MTO; PA_MTO (Other Grant/Funding Number: Changi General Hospital)
Record Dates: First submitted 2023-10-13; First posted 2023-10-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Primary Aldosteronism Due to Aldosterone Producing Adenoma; Primary Aldosteronism; Adrenal Tumors
Keywords: 11-C Metomidate PET/CT; Functional imaging; Secondary / Endocrine hypertension; Adrenal Vein Sampling; Subtyping; localization testing; Adrenalectomy
MeSH Terms: conditions — Hyperaldosteronism; Adrenal Gland Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: 11C-metomidate synthesis will be done at Clinical Imaging Research Centre in compliance with good manufacturing practice using a General Electric Medical Systems PET trace 860 cyclotron. Non-contrast CT images will be acquired over the adrenal. After an intravenous injection of 11C-metomidate, PET images will be acquired. Attenuation and decay-corrected images will be converted to standardized uptake value (SUV) maps through division by (injected activity per patient weight). The maximum SUV values over regions of interest will be determined for 10-min static images starting 35 min after the injection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 11C-metomidate PET-CT (Experimental): All patients will undergo standard-of-care investigations (CT imaging of adrenals and AVS) and the research test (11C-metomidate PET-CT) with a dose of 100 - 300 Megabecquerel (MBq) (11C-metomidate) to identify functional unilateral adrenal disease
  Interventions: Combination Product: 11C-Metomidate PET/CT imaging at Clinical Imaging Research Centre

INTERVENTIONS:
Combination Product: 11C-Metomidate PET/CT imaging at Clinical Imaging Research Centre — 11C-Metomidate PET/CT imaging at Clinical Imaging Research Centre

SUMMARY:
* 10% of patients with hypertension potentially have the treatable condition - primary aldosteronism (PA). This is caused by either bilateral adrenal disease (~40%), managed with lifelong medications; or unilateral disease (~60%), cured with laparoscopic surgery (adrenalectomy). Current diagnosis of PA includes a screening test with aldosterone-renin ratio, followed by a confirmatory salt loading test (in most patients) to demonstrate unsuppressed aldosterone levels. Of note, some patients with suppressed aldosterone after confirmatory tests (also termed low-renin hypertension) may also have unilateral adrenal tumors.
* The difficulty with identifying curable unilateral disease is due to adrenal vein sampling (AVS): an invasive, and technically-difficult procedure. An alternative novel imaging, 11C-Metomidate Positron emission tomography-computed tomography (PET-CT), can detect adrenal tumors which are over-producing aldosterone. It is non-invasive, non-operator-dependent, and potentially may identify more patients with curable unilateral disease. The results from our pilot study in 25 patients with confirmed PA (ClinicalTrials.gov NCT03990701, PA_CURE) showed that 11C-Metomidate PET-CT exhibited comparable performance to AVS in subtyping PA, and this should be validated in a larger study.
* In addition, 11C-Metomidate is also able to differentiate adrenocortical lesions in the adrenal gland from other lesions found in adrenal tissue, such as adrenomedullary lesions (e.g. pheochromocytoma).
* Hence, the investigators hypothesize that 11C-metomidate PET-CT can accurately (1) identify patients with surgically curable unilateral adrenal disease among hypertensive Asians with primary aldosteronism (PA_CURE 2 / PA_MTO EH study) and (2) differentiate adrenocortical lesions from other lesions in patients with adrenal tumors (PA_MTO AT study)

DETAILED DESCRIPTION:
* The investigators aim to recruit 100 patients with confirmed, or likely, primary aldosteronism to undergo conventional tests, CT, AVS, and 11C-metomidate PET-CT.
* Results will be reviewed and discussed at a multidisciplinary meeting, and patients with unilateral PA or adrenal tumor will be offered surgery. Patients will be reviewed 6 months post-surgery.
* In a separate study, the investigators will recruit 10 patients with adrenal tumors to differentiate adrenocortical lesions from other lesions in patients with adrenal tumors

ELIGIBILITY:
Inclusion Criteria:

* For patients with primary aldosteronism (PA_CURE 2 / PA_MTO EH):

  1. Confirmed diagnosis of primary aldosteronism, as defined in Endocrine Society Guidelines 2016, with positive confirmatory test (post-salt loading aldosterone >140pmol/L); or hypokalemia with undetectable renin levels and aldosterone >550pmol/L; or likely primary aldosteronism / low-renin hypertension (inappropriate aldosterone levels and suppressed renin levels)
  2. Keen for surgical treatment if shown to have unilateral adrenal disease.
* For patients with suspected adrenal tumors (PA_MTO AT)

  1. All patients with suspected adrenal tumors based on imaging and clinical suspicion.

Exclusion Criteria:

* Inability to provide written informed consent.
* Chronic renal failure of Stage 3b or greater severity, estimated glomerular filtration rate (eGFR) < 45ml/min/1.73m2 using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula. (only applicable for PA_CURE 2 / PA_MTO EH)
* Severe or terminal medical condition(s) that in the view of the investigator prohibits participation in the study or interferes with possible treatment or health-related quality of life, e.g. cancer, end-stage liver disease, end stage renal failure (only applicable for PA_CURE 2 / PA_MTO EH)
* Contraindications to isotope scanning (e.g. Female patients who are pregnant (self-declared or via positive pregnancy test), intending to become pregnant (within 3 months of scan) or breastfeeding) or CT Scan, which includes but not limited to waist circumference >140cm, morbid obesity or claustrophobia (limiting entry in CT scanner)
* Contraindication to ingestion of corticosteroids (e.g. poorly controlled diabetes, HbA1C >13%)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-12-30 (Actual); Primary Completion 2025-05-25 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Biochemical outcome of unilateral primary aldosteronism based on the Primary Aldosteronism Surgical Outcome (PASO) criteria (PA_CURE 2 / PA_MTO EH study). | 6 months
  The number of patients with complete, partial, and absent biochemical success according to the PASO criteria.
Diagnostic performance of 11C-Metomidate PET-CT in identifying unilateral adrenocortical tumor (PA_MTO AT study). | 6 months
  Percentage of patients accurately identified with adrenocortical tumor using 11C-Metomidate PET-CT, when compared to the histopathology of the excised tumor. In patients who have not undergone surgery, this will be determined by clinical diagnosis.

SECONDARY OUTCOMES:
Clinical outcome of unilateral primary aldosteronism based on the Primary Aldosteronism Surgical Outcome (PASO) criteria (PA_CURE 2 / PA_MTO EH STUDY). | 6 months
  The number of patients with complete, partial, and absent clinical success according to the PASO criteria.
Diagnostic performance of 11C-Metomidate PET-CT in identifying unilateral aldosterone-producing adenoma (PA_CURE 2 / PA_MTO EH study). | 6 months
  Percentage of patients accurately identified with unilateral PA using 11C-Metomidate PET-CT and AVS, as compared to histopathology of the excised tumor (defined as 'Classical' single, functioning aldosterone-producing adenoma using HISTopathological classification by the Histopathology of primary ALDOsteronism (HISTALDO) consensus).
Cost-effectiveness of 11C-Metomidate PET-CT versus AVS in diagnosing patients with unilateral primary aldosteronism (PA_CURE 2 / PA_MTO EH STUDY). | 6 months
  Cost-effectiveness of the diagnostic course will be calculated by using calculated costs per quality-adjusted life years (QALYs).
Diagnostic criteria using 11C-metomidate PET/CT (PA_CURE 2 / PA_MTO EH study). | 6 months
  The cut-off level of maximum standard update value (SUVmax) values which offer the best sensitivity and specificity for lateralization of aldosterone-producing adenoma in 11C-metomidate PET/CT.
Number of patients with low-renin hypertension with unilateral adrenal tumors (PA_CURE 2 / PA_MTO EH study). | 6 months
  Quantify the number of patients with low-renin hypertension or only obtain borderline diagnostic criteria for PA but have unilateral adrenal lesions detected on 11C-metomidate PET/CT.

CONTACTS AND LOCATIONS:
Locations (7):
- Singapore (7):
  - Changi General Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore
  - National University Hospital, Singapore
  - Ng Teng Fong General Hospital, Singapore
  - Sengkang General Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No